CLINICAL TRIAL: NCT04383392
Title: A Cross-over Randomized Controlled Trial of Quality of Life Between Cardiovascular Implantable Electronic Device With and Without Rate Adaptive Pacing
Brief Title: QoL Between CIEDs With and Without Rate Adaptive Pacing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NTUHHsin-Chu
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Pacemaker DDD; Quality of Life
Keywords: rate adaptive; pacemaker; quality of life

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rate adaptive pacing (Experimental): Turn on Rate adaptive pacing
  Interventions: Device: Rate adaptive pacing
- No Rate adaptive pacing (Active Comparator): Turn off Rate adaptive pacing
  Interventions: Device: Rate adaptive pacing

INTERVENTIONS:
Device: Rate adaptive pacing — Rate-adaptive pacing is a function of permanent pacemaker to accelerate patients' heart rate when they are walking, stair climbing, running or carrying on intensive physical activity. Appropriately, the function is similar to human's electrophysiology of sinus node but it may be difficult to replace sinus node's function totally. For example, the acceleration or deceleration slope when exercise beginning or cessation is not always the same or consistent in different patients and different time.

SUMMARY:
Clinical implantable electronic devices, such as permanent pacemaker, implantable cardioverter defibrillator and cardiac resynchronization therapy are used in current daily practice for patients with bradycardia, ventricular arrhythmia, or heart failure. The rapid progress of permanent pacemaker function is growing to replace human's degenerating electrophysiology of heart.

The ability of physical work is an important cornerstone of quality of life. In daily activities, rate response to higher rate is importance for patients with bradycardia who can not accelerate their heart rate. And rate-adapting pacing of permanent pacemaker is a design to increase heart rate pacing according to physical activity or emotional activity. Patients with rate-adaptive pacing will get more cardiac output and overcome the physical activity such as stair climbing. But there are few studies to evaluate whether the rate-adaptive pacing of permanent pacemaker will improve the quality of life in people with bradycardia. The aim of this study is to compare turn-on with turn-off this function (DDDR vs DDD) whether rate-adaptive pacing will improve quality of life in patients with permanent pacemakers.

ELIGIBILITY:
Inclusion Criteria:

* sick sinus syndrome for permanent dual-chamber pacing
* pacemakers are implanted for ≥30 days with no complications.

Exclusion Criteria:

* (1) patient or legal representative could not provide written informed consent
* (2) unwillingness or inability to return for follow-up visits or reason to believe that adherence to follow-up visits wound be irregular,
* (3) current or scheduled enrollment in other, conflicting studies,
* (4) concomitant disease or other medical condition likely to result in death within 6 months, and

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Short-Form 36 Questionnaire | 3 months
  The SF-36 questionnaire consists of eight health concepts (1) physical functioning, (2) role limitations due to physical health, (3) bodily pain, (4) general health perceptions, (5) vitality (energy/fatigue), (6) social functioning, (7) role limitations due to emotional health, (8) general mental health (psychological distress/wellbeing) which are expressed as a score on a 0-100 scale for each of the eight health concepts. The maximum score of 100 means no disability in five of the scales (Physical Functioning, Role Physical, Bodily Pain, Social Functioning, and Role Emotional) and indicates not the absence of disability, but the presence of a positive state of health in the other scales (General Health, Vitality and Mental Health).

SECONDARY OUTCOMES:
6 minute walking test | 3 months
NYHA functional class | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Hsinchu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No